CLINICAL TRIAL: NCT06446076
Title: Feedback Using behaviOral econOmic Theories on STEP countS in Cardiovascular Disease Patients: A Randomized Controlled Trial
Brief Title: Feedback Using behaviOral econOmic Theories on STEP countS in Cardiovascular Disease Patients
Acronym: FOOTSTEPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's International Hospital, Japan (Other)
Collaborators: Trigen (Industry)
Responsible Party: Principal Investigator, Atsushi Mizuno, Director, Medical quality management office, St. Luke's International Hospital, Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-RCK043
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Rehabilitation; Behavioral Economics
Keywords: Cardiovascular diseases; Rehabilitation; Behavioral Economics; Health Services
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control group (No Intervention): Participants in this group will not receive goal-setting or gamification interventions during the 6-week intervention period and the additional 6-week follow-up period. As an "active control" during the 12-week trial period, participants will be able to check their daily step counts using an application with the same specifications.
- Gamification (Loss framing) (Experimental): This group will receive a gamification intervention with loss framing.
  Interventions: Behavioral: Gamification (Gain/Loss framing)
- Gamification (Gain framing) (Experimental): This group will receive a gamification intervention with gain framing.
  Interventions: Behavioral: Gamification (Gain/Loss framing)
- Gamification (Loss framing) + Social support (Experimental): This group will receive a gamification intervention with loss framing and a social support intervention.
  Interventions: Behavioral: Gamification (Gain/Loss framing); Behavioral: Social support
- Gamification (Gain framing) + Social support (Experimental): This group will receive a gamification intervention with gain framing and a social support intervention.
  Interventions: Behavioral: Gamification (Gain/Loss framing); Behavioral: Social support

INTERVENTIONS:
Behavioral: Gamification (Gain/Loss framing) — Participants will take part in a 6-week game-based program designed to help them reach their daily step goals. They are encouraged to maintain their daily step counts to achieve their daily step target over the 6-week intervention period. The gamification design incorporates two theoretically effective behavioral economics principles, "Fresh Start" and "Loss Aversion". All participants start from the Silver rank (middle rank), and their rank changes based on each final point of the week. The ranks are set from top to bottom as Platinum, Gold, Silver, Bronze, and Blue. In loss framing, if the daily step target is 6000 steps, maintaining 70 points for achieving 6000 steps on day 1, and a deduction of 10 points for not achieving it. In gain framing, achieving 6000 steps on day 1 results in an addition of 10 points, with no increase for not achieving it. After one week, ranks increase if the points at midnight on Sunday are 40 or above, and decrease if below this threshold.
  Arms: Gamification (Gain framing); Gamification (Gain framing) + Social support; Gamification (Loss framing); Gamification (Loss framing) + Social support
Behavioral: Social support — Participants in this group are asked to designate a family member or friend to provide social support. This supporter is encouraged to check the participant's progress and provide support during the interventional period. The supporter will also receive weekly emails throughout the period, informing them about the participant's daily step counts, achievement status, points, levels, and other relevant information.
  Arms: Gamification (Gain framing) + Social support; Gamification (Loss framing) + Social support

SUMMARY:
This is a prospective, randomized controlled trial. The aim of the study is to verify the effectiveness of interventions using gamification with social incentives and social support to increase physical activity in patients with CVD through randomized controlled trials.

DETAILED DESCRIPTION:
The three aims of this randomized controlled trials;

1. To demonstrate the effectiveness of loss framing in gamification for achieving increased physical activity in patients with CVD.
2. To demonstrate the effectiveness of social support in gamification for achieving increased physical activity in patients with CVD.
3. To evaluate the impact of the intervention using social incentives and social support through gamification on changes in participants; subjective assessment of physical activity levels, body mass index (BMI), and lipid panel in blood tests.

Secondary Objective:

1. To assess whether the differences between study groups in achieving the goal of increased physical activity during the 6-week intervention period persist during the 6-week follow-up period.
2. To investigate how the increase in physical activity through gamification in patients with CVD is influenced by patients; behavioral characteristics and environmental factors.

This trial will be a five-group, randomized controlled trial (RCT) with an intervention period of 6 weeks and a follow-up period of additional 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of old myocardial infarction or chronic heart failure
* Ability to read and provide informed consent to participate in this trial
* Owning a smartphone capable of installing this application

Exclusion Criteria:

* Having difficulty using smartphones (due to vision problems or IT literacy issues)
* Exercise therapy is contraindicated (in accordance with the 2021 revised guidelines on rehabilitation in cardiovascular diseases)
* Ability to read and provide informed consent to participate in this trial
* Owning a smartphone capable of installing this application
* Participating in other studies related to physical activity
* Being pregnant
* Any other medical conditions or reasons they are unable to participate in a physical activity study for 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean daily step counts | From enrollment to the end of intervention period at 8 weeks (2-weeks run-in and 6-weeks intervention period)
  The primary outcome is change in mean daily step counts from baseline to the 6-week intervention period.

SECONDARY OUTCOMES:
Percentage of days achieving their step goals | From enrollment to the end of follow-up period at 14 weeks
  Secondary outcomes include the percentage of days achieving their step goals during the intervention and follow-up periods and the change in daily step counts from baseline to follow-up period.

OTHER OUTCOMES:
Change in International Physical Activity Questionnaire (IPAQ) | From enrollment to the end of follow-up period at 14 weeks
  Change in the participant's subjective assessment of physical activity level measured using the International Physical Activity Questionnaire (IPAQ) Short Form. This is a survey that investigates how individuals engage in physical activity (how they move their bodies) in their daily lives. It is a questionnaire that assesses the duration and frequency of exercise based on intensity levels.
Change in Body weight (BMI) | From enrollment to the end of follow-up period at 14 weeks
  Change in body weight (BMI) (kg/m^2)
Change in LDL/HDL cholesterol | From enrollment to the end of follow-up period at 14 weeks
  Change in LDL/HDL cholesterol (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Mizuno, MD, PhD, Principal Investigator — Department of Cardiovascular Medicine, St. Luke's International Hospital
Locations (1):
- St. Luke's International Hospital, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suzuki T, Aoki J, Abe K, Asano T, Yoneoka D, Sato S, Rewley J, Miyata K, Ono M, Saito A, Kanie T, Okui K, Takahashi A, Isa K, Takasago S, Shiina Y, Nishihata Y, Niinuma H, Masuda K, Kijima Y, Nishida H, Komiyama N, Sugibuchi K, Suzuki Y, Igarashi A, Suzumura S, Tsurugi N, Okamura D, Mizuno A; FOOTSTEPS Investigators. Rationale and Trial Design of Feedbacks Using Behavioural Economic Theories on STEP Counts (FOOTSTEPS) Trial in Patients With Cardiovascular Disease. CJC Open. 2024 Dec 27;7(4):535-544. doi: 10.1016/j.cjco.2024.12.009. eCollection 2025 Apr. PMID 40433138